CLINICAL TRIAL: NCT07114068
Title: Does Self-Soft Tissue Mobilization of Obturator Internus Reduce Pelvic Floor or Hip Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Fox University (Other)
Responsible Party: Principal Investigator, Tess Treinen Swake, Physical Therapist, Assistant Professor, George Fox University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2231085
Record Dates: First submitted 2025-08-03; First posted 2025-08-11 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Pelvic Floor Dysfunction; Hip Pain
Keywords: self soft tissue mobilization; pelvic floor dysfunction; active females

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internal Mobilization Group (Active Comparator): This group performs self mobilization of the Obturator Internus muscle internally.
  Interventions: Other: Self mobilization of Obturator Internus Muscle using wand
- External Mobilization Group (Active Comparator): This group performs self mobilization of the Obturator Internus muscle externally.
  Interventions: Other: Self mobilization of Obturator Internus Muscle using wand

INTERVENTIONS:
Other: Self mobilization of Obturator Internus Muscle using wand — Participants will be randomly assigned to the internal or external Obturator Internus mobilization groups. The internal mobilization group will access the Obturator Internus muscle via the vagina, which is common practice in Pelvic Health Physical Therapy. The external mobilization group will be accessing the Obturator Internus muscle with the same pelvic wand, but externally. Pelvic wands will be provided for each participant at no cost and will be used for only that participant. Prior to intervention with a pelvic wand, each participant will be provided education regarding the anatomy of the pelvic floor and hip and a protocol review of the intervention.

SUMMARY:
The Obturator Internus is a muscle deep within the pelvis. Fifty percent of the muscle belly can be palpated internally within the pelvic floor and 50% of the muscle externally in the pelvis. This muscle is unique in the sense that it is both a muscle of the pelvic floor as well as a muscle of the hip. There is limited research for addressing Obturator Internus muscle dysfunction in rehabilitation, but during specialty training in Pelvic Health Physical Therapy, manual techniques addressing Obturator Internus tension are indicated as a treatment to reduce dysfunction with soft tissue mobilization. The goal of this research is twofold. Firstly, to assess if self-soft tissue mobilization of the Obturator Internus muscle is beneficial for active females with pelvic floor relaxing or nonrelaxing dysfunction (PFD) or hip pain, and secondly if internal or external mobilization of the Obturator Internus muscle is more beneficial.

DETAILED DESCRIPTION:
The objectives of this study are to assess if self-soft tissue mobilization of the Obturator Internus muscle with a pelvic wand reduces relaxing or nonrelaxing PDF or hip pain and if symptoms are reduced, which group experienced a greater improvement (internal or external Obturator Internus mobilization). Participants will be randomly assigned to the internal or external Obturator Internus mobilization groups. The internal mobilization group will access the Obturator Internus muscle via the vagina, which is common practice in Pelvic Health Physical Therapy. The external mobilization group will be accessing the Obturator Internus muscle with the same pelvic wand, but externally. Pelvic wands will be provided for each participant at no cost and will be used for only that participant. Prior to intervention with a pelvic wand, each participant will be provided education regarding the anatomy of the pelvic floor and hip and a protocol review of the intervention. There will be initial data collected prior to beginning self-soft tissue mobilization, data collected at a midpoint and following the intervention protocol. Data will be collected via a survey in REDCap (HIPAA-compliant), created specifically for this research, which includes demographics, injury history, history of PFD and/or hip pain, characteristics of physical activity and/or sport(s), knowledge of pelvic floor musculature, and questions regarding the correlation between PFD and performance. International Consensus on Incontinence Questionnaire (ICIQ-FLUTS Long Form) and Patient Reported Outcomes Measurement Information System (PROMIS) questions to address biopsychosocial concerns (specifically Anxiety & Depression) are also included.

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-45 years
* Female gender
* Current pelvic floor dysfunction (relaxing or nonrelaxing) or current hip pain
* Participants must be physically active as defined by the World Health Organization as performing 150-300 minutes of moderate-intensity aerobic physical activity or at least 75-150 minutes of vigorous-intensity aerobic physical activity; or an equivalent combination of moderate- and vigorous-intensity activity throughout the week.

Exclusion Criteria:

* Pregnancy
* Gynecological or Obstetric Surgery within 6 months
* Active infection (including Sexually Transmitted Infection, Pelvic, Yeast)
* Cancer
* Inflammatory Disease
* Connective Tissue Disease
* Or have been instructed by a Healthcare provider to not participate

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-01-28 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-05-27 (Actual)

PRIMARY OUTCOMES:
International Consensus on Incontinence Questionnaire (ICIQ-FLUTS Long Form) | At enrollment and completion (2 weeks later)
  A questionnaire that evaluates female lower urinary tract symptoms and quality of life in clinical practice and research. This questionnaire has been found to be valid, reliable, and responsive.
Patient Reported Outcome Measure Information System (PROMIS): Anxiety & Depression | Initial enrollment and at completion (2 weeks later)
  measures are scored on the T-score metric. Higher scores mean more of the attribute being measured (e.g., more Fatigue, more Physical Function). Thus, a score of 60 is one standard deviation above the average reference population. PROMIS measures are rigorously developed and validated self-report tools spanning 300+ measures across physical, mental, and social health (https://www.healthmeasures.net/explore-measurement-systems/promis/intro-to-promis). As a Computer Adaptive Test (CAT), each measure asks 4-10 questions (average 5-6) drawn from the total item bank.

CONTACTS AND LOCATIONS:
Locations (1):
- George Fox University Medical Sciences Building, Newberg, Oregon, United States

REFERENCES:
- [Background] Muro S, Nimura A, Ibara T, Chikazawa K, Nakazawa M, Akita K. Anatomical basis for contribution of hip joint motion by the obturator internus to defaecation/urinary functions by the levator ani via the obturator fascia. J Anat. 2023 Apr;242(4):657-665. doi: 10.1111/joa.13810. Epub 2022 Dec 18. PMID 36528838
- [Background] Morris VC, Murray MP, Delancey JO, Ashton-Miller JA. A comparison of the effect of age on levator ani and obturator internus muscle cross-sectional areas and volumes in nulliparous women. Neurourol Urodyn. 2012 Apr;31(4):481-6. doi: 10.1002/nau.21208. Epub 2012 Feb 29. PMID 22378544
- [Background] Meister MR, Sutcliffe S, Ghetti C, Chu CM, Spitznagle TM, Lowder JL. A pilot trial of movement-based pelvic floor physical therapy to address pelvic floor myofascial pain and lower urinary tract symptoms. Int Urogynecol J. 2023 Jun;34(6):1261-1270. doi: 10.1007/s00192-022-05353-9. Epub 2022 Sep 20. PMID 36125508
- [Background] Lewis GK, Chen AH, Craver EC, Crook JE, Carrubba AR. Trigger point injections followed by immediate myofascial release in the treatment of pelvic floor tension myalgia. Arch Gynecol Obstet. 2023 Apr;307(4):1027-1035. doi: 10.1007/s00404-022-06880-y. Epub 2022 Dec 14. PMID 36513896
- [Background] Crowle, A., and C. Harley. "Exploration of the Efficacy of Myofascial Release and Trigger Point Therapy for Women with Pelvic Organ Prolapse." Physiotherapy 107 (2020): e104-e104. Web.
- [Background] Cage, Stephen A., and Brandon J. Warner. "Idiopathic Obturator Internus Strain in a Collegiate Tennis Player: A Case Report." The Journal of Sports Medicine and Allied Health Sciences 3.2 (2017): n. pag. Web.
- [Background] Anderson RU, Wise D, Sawyer T, Nathanson BH, Nevin Smith J. Equal Improvement in Men and Women in the Treatment of Urologic Chronic Pelvic Pain Syndrome Using a Multi-modal Protocol with an Internal Myofascial Trigger Point Wand. Appl Psychophysiol Biofeedback. 2016 Jun;41(2):215-24. doi: 10.1007/s10484-015-9325-6. PMID 26721470
- [Background] Anderson R, Wise D, Sawyer T, Nathanson BH. Safety and effectiveness of an internal pelvic myofascial trigger point wand for urologic chronic pelvic pain syndrome. Clin J Pain. 2011 Nov-Dec;27(9):764-8. doi: 10.1097/AJP.0b013e31821dbd76. PMID 21613956